CLINICAL TRIAL: NCT00346528
Title: Safety of NGOIS Compared to BSS Plus in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-64
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — glutathione-bicarbonate-Ringer solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NGOIS (Experimental)
  Interventions: Drug: Next Generation Ophthalmic Irrigating Solution (NGOIS)
- BSS Plus (Active Comparator)
  Interventions: Drug: BSS Plus

INTERVENTIONS:
Drug: Next Generation Ophthalmic Irrigating Solution (NGOIS) — Volume sufficient to irrigate adequately during cataract surgery
  Arms: NGOIS
Drug: BSS Plus — Volume sufficient to irrigate adequately during cataract surgery
  Arms: BSS Plus

SUMMARY:
To evaluate the Safety of Next Generation Ophthalmic Irrigating Solution compared to BSS Plus for use during cataract surgery in Pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Cataract present.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* As per age requirements.
* Other protocol-defined exclusion criteria may apply.

Ages: 1 Week to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety Variables: Endothelial cell density, visual acuity, intraocular pressure, ocular signs and fundus assessment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lane, Study Director — Medical Monitor
Locations (1):
- Contact Alcon for Trial Locations, Fort Worth, Texas, United States